CLINICAL TRIAL: NCT07165405
Title: The Effect of Hot Sacral Massage With Cherry Pits and Shower Application With Partner Support on Perceived Labor Pain, Birth Experience, and Birth Comfort
Brief Title: Effects of Hot Sacral Massage and Shower Application With Partner Support on Labor
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Neriman Guducu, Assistant Professor, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 12/32
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Pain; Experience; Comfort
Keywords: labor pain; birth experience; postpartum comfort; sacral massage; shower application
MeSH Terms: conditions — Pain; Labor Pain | interventions — Massage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Showering with Partner Support (Experimental): Participants in this group will receive a shower administered by their partner on their back, abdomen, or entire body while standing or sitting, with the water temperature maintained between 32-37°C (the woman's preferred temperature will be applied) for at least 20 minutes upon admission to the labor room (when dilation is 4-5 cm). This will be performed under the observation of the researcher midwife. The application will be repeated when dilation reaches 7-8 cm.
  Interventions: Other: Shower
- Hot Sacral Massage Group Made with Cherry Pits (Experimental): Sacral Massage Application will be performed using 20x20 cm pouches filled with cherry pits. Like the shower application, massage will be performed upon admission to the delivery room (when dilation is 4-5 cm) and repeated when dilation reaches 7-8 cm. Unless the pregnant woman requests otherwise, massage will be performed while she is in the left lateral position.
  Interventions: Other: Massage
- Control Group (Other): Participants in this group will not receive any treatment beyond the routine hospital protocol (midwifery care).
  Interventions: Other: Midwifery Care

INTERVENTIONS:
Other: Shower — Participants in this group will receive a shower administered by their partner on their back, abdomen, or entire body while standing or sitting, with the water temperature maintained between 32-37°C (the woman's preferred temperature will be applied) for at least 20 minutes upon admission to the labor room (when dilation is 4-5 cm). This will be performed under the observation of the researcher midwife. The application will be repeated when dilation reaches 7-8 cm.
  Arms: Showering with Partner Support
Other: Massage — Sacral Massage Application will be performed using 20x20 cm pouches filled with cherry pits. Like the shower application, massage will be performed upon admission to the delivery room (when dilation is 4-5 cm) and repeated when dilation reaches 7-8 cm. Unless the pregnant woman requests otherwise, massage will be performed while she is in the left lateral position.
  Arms: Hot Sacral Massage Group Made with Cherry Pits
Other: Midwifery Care — Care provided by a midwife in the delivery room
  Arms: Control Group

SUMMARY:
This study was designed to determine the effect of warm sacral massage with cherry pits and showering with partner support on perceived labor pain, birth experience, and birth comfort. A total of 150 pregnant women, 50 in each group, were planned to be included in the study.

Volunteers who agreed to participate in the study were expected to have spontaneous vaginal delivery, with an ultrasound-estimated fetal weight between 2500-4000 grams, a single fetus in cephalic presentation, at term (between 37-42 weeks of gestation), in the active phase of labor (4 cm cervical dilation), primiparous women who did not receive analgesia or anesthesia during the first stage of labor and who did not have any skin disease or open wound that would prevent massage or showering. Pregnant women participating in the study will be randomly divided into three groups. The massage group will receive massage twice during the first stage of labor for at least 20 minutes, either standing or sitting, using a bag filled with cherry pits on the sacral region (the lumbar region including your tailbone). Pregnant women in the shower group will receive a shower with water at a temperature between 32-37°C for at least 20 minutes twice during the first stage of labor, either standing or sitting with partner support, according to their preference. Pregnant women in the control group will not receive any intervention other than the routine hospital protocol (midwifery care).

After providing information about the study to the pregnant women, written informed consent will be obtained. The pain scale (VAS) will be administered to women in the shower group, massage group, and control group by a midwife working in the delivery room who is not involved in the study. The VAS will be administered four times during labor to pregnant women in the massage group and shower group, and four times to pregnant women in the control group.

Before transfer to the ward after delivery, all participants in the groups will be administered the "Birth Experience Scale (BES) and Birth Comfort Scale (BCS)" by a midwife who is not involved in the study and is working in the delivery room that day.

DETAILED DESCRIPTION:
This study aims to determine the effect of warm sacral massage with cherry pits and shower application with partner support on perceived labor pain, birth experience, and birth comfort. The study includes three groups: massage group, shower group, and control group. A total of 150 pregnant women, 50 in each group, were included in the study.

Steps for the Partner-Assisted Shower Application: Participants in this group will receive a shower administered by their partner in the delivery room (when dilation is 4-5 cm) for at least 20 minutes. The water temperature will be between 32-37 °C (the woman's preferred temperature will be used), and the shower will be administered to the lower back, abdomen, or entire body, depending on the woman's preference, while she is standing or sitting, under the observation of the researcher midwife. The application will be repeated when dilation reaches 7-8 cm. To ensure the safety of pregnant women before showering, non-slip sandals or slippers will be provided, and a non-slip bath mat will be placed under the stool. Blood pressure will be checked before and after showering.

Cherry Pit Hot Sacral Massage Group: The sacral massage will be performed using 20x20 cm pouches filled with cherry pits. The pouches will be cover-shaped, and 100% cotton fabric will be preferred. Each pregnant woman will receive a massage with a washed, clean pouch. Like the shower application, the massage will be performed upon admission to the delivery room (when dilation is 4-5 cm) and repeated when dilation is 7-8 cm. It will begin when contractions start and will last approximately 20 minutes.

Control group application steps: Participants in this group will not receive any application other than the routine hospital protocol (midwifery care).

The vital signs (blood pressure, pulse) of all pregnant women in the groups will be measured hourly by the midwife and recorded in each participant's file.

The VAS will be administered to women in the shower group, massage group, and control groups by a midwife working in the delivery room who is not involved in the study. The VAS will be measured four times during the first stage of labor for pregnant women in the shower and massage groups.

After delivery, before transfer to the ward, the "Birth Experience Scale (BES) and Birth Comfort Scale (BCS)" will be administered to all participants in the groups by a midwife who is not involved in the study and who is working in the delivery room that day.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Expectation of spontaneous vaginal delivery
* Estimated fetal weight between 2500-4000 grams by ultrasound
* Single fetus and cephalic presentation,
* Term pregnancy (between 37-42 weeks of gestation)
* Being in the active phase of labor (cervical dilation of 4 cm)
* No analgesia or anesthesia used during the first stage of labor,
* No skin disease or open wound preventing massage or showering

Exclusion Criteria:

* Having undergone infertility treatment,
* Delivery by cesarean section for any reason during labor,
* Being multiparous
* Having any systemic, chronic, or neurological disease (Diabetes Mellitus, Hypertension, Thyroid disorders, Multiple Sclerosis, Epilepsy, etc.)
* Regular medication use due to any illness,
* Active psychiatric treatment (pharmacotherapy/psychotherapy),
* Any induction that may affect uterine contractions and dilation,
* Any pregnancy complications (such as placenta previa, preeclampsia, premature rupture of membranes, oligohydramnios, and polyhydramnios)
* Interventional delivery (forceps, vacuum)
* Any problem that hinders communication (such as not knowing Turkish, hearing, speech, and comprehension disorders)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 150 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
visual analog scale | Before the shower and massage at 4-5 cm dilation, After the shower and massage at 4-5 cm dilation, Before the shower and massage at 6-8 cm dilation, After the shower and massage at 6-8 cm dilation. Control group: at 4-5 cm dilation and 6-8 cm dilation
  labour pain

SECONDARY OUTCOMES:
Childbirth Experience Questionnaire | Before the transfer from the delivery room to the maternity ward after birth
  The scale to be used to measure women's birth experiences in different dimensions has four sub-dimensions and 22 items. In the birth process sub-dimension, women's sense of personal control and their feelings about the birth process and birth pain are evaluated. In the professional help/support sub-dimension, information and midwifery care are evaluated. The perceived safety/memories sub-dimension examines feelings of safety and memories/records of the birth. The participation in decisions sub-dimension examines participation in decisions regarding movement, birth position, and pain relief. A higher score on the scale indicates that the expectant mother had a positive birth experience.
Childbirth Comfort Questionnaire | Before the transfer from the delivery room to the maternity ward after birth
  The scale has a 3-factor structure (physical, environmental, psychospiritual). It is used to assess the woman's comfort level during childbirth. A higher score indicates a higher level of comfort, while a lower score indicates a lower level of comfort.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpaşa, Istanbul, Büyükçekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No